CLINICAL TRIAL: NCT03379168
Title: Evaluating the Efficacy of Micro-fragmented Adipose Tissue and Intra-articular Corticosteroid Injections for Symptomatic Knee Osteoarthritis: a Randomized, Placebo Controlled Study.
Brief Title: Efficacy of Micro-fragmented Adipose Tissue Injection for Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dustin L. Richter, MD (Other)
Responsible Party: Sponsor-Investigator, Dustin L. Richter, MD, Assistant Professor, Department Orthopaedic Surgery, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-146
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; mesenchymal stem cell; adipose tissue; injection; nonoperative treatment
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized, placebo-controlled clinical trial. Patients will be randomized to receive either Lipogems, intra-articular corticosteroids, or a placebo injection of saline. Lipogems is cleared for use by the FDA in orthopaedics and arthroscopy and is offered as a treatment option for knee osteoarthritis. This study will be evaluating the effectiveness (not safety) of Lipogems when compared to corticosteroids and placebo. Thus, no information will be submitted to the FDA.
Who Masked: Participant
Masking Description: It is not feasible to blind patients who are randomized to receive Lipogems, as adipose tissue must be obtained from the participant. However, patients randomized to receive intra-articular corticosteroids or placebo injections will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Placebo Injection (Placebo Comparator): Patients who are randomized to the placebo group will receive an injection of 7cc of sterile saline in the affected knee.
  Interventions: Drug: Saline
- Corticosteroid Injection (Active Comparator): Patients who are randomized to the corticosteroid group will receive an injection of 2cc (80mg) of triamcinalone acetonide injectable suspension mixed with 5 cc of 1% plain lidocaine for a total of 7cc of fluid injected in the affected knee.
  Interventions: Drug: Corticosteroid injection
- Lipogems Injection (Experimental): Patients who are randomized to the Lipogems treatment group will undergo a lipoaspiration from their abdomen and autologous injection of the harvested adipocytes into their knee. It is standard to harvest three to four times more adipose tissue than is planned to be injected to account for tissue processing by the Lipogems device. The investigators plan to inject 7cc of autologous adipose tissue. Thus, the investigators will harvest between 25 and 30 cc of adipose tissue from each patient. The tissue will be processed immediately and 7cc will be injected. Any remaining adipose tissue will be disposed of immediately in biohazardous waste.
  Interventions: Device: Microfragmented Adipose Tissue (Lipogems)

INTERVENTIONS:
Device: Microfragmented Adipose Tissue (Lipogems) — Lipogems is a technique to harvest, process, and inject minimally manipulated adipose tissue. This procedure is enzyme free and requires no clonal expansion or manipulation. Lipoaspirate is harvested most commonly from the abdomen and washed in saline solution, then processed through a closed-system device that micro-fragments the adipose tissue. This mechanical process retains the vascular architecture, mature pericytes, and MSCs for autologous injection. Lipogems is currently FDA-approved for orthopedic and arthroscopic procedures; thus, this would be an on-label use for knee injections.
  Arms: Lipogems Injection
Drug: Corticosteroid injection — Cortisone is a standard of care injection to reduce joint inflammation.
  Arms: Corticosteroid Injection
Drug: Saline — Sterile saline injection will act as a placebo group.
  Arms: Placebo Injection

SUMMARY:
Knee osteoarthritis (OA) causes patients considerable joint pain and leads to instability, reduced range of motion, and functional limitations. Current treatment limitations have generated interest in alternative options to restore function and alleviate joint pain, some with the aim of healing damaged articular cartilage. There has been preliminary support in the literature for reduced pain and improved functional performance in patients who receive mesenchymal stem cells (MSCs) as part of a treatment regimen. MSCs can be costly and are limited by complex regulatory issues. This interest in an alternative isolation method lead to the development of Lipogems. Lipogems is a technique to harvest, process, and inject minimally manipulated adipose tissue. This procedure is enzyme free and requires no clonal expansion or manipulation. The goal of this study is to evaluate the possible benefits of reduced joint pain and increased joint functionality in patients with knee osteoarthritis after the injection of Lipogems. In addition, given the limitations of prior research on the efficacy of intra-articular corticosteroids, the investigators will also include this as an additional study group to compare to placebo. There have been case reports published showing favorable outcomes. This would be the first study reporting data on the efficacy of Lipogems for pain relief in knee OA in a randomized, controlled clinical trial with a larger sample of patients.

The investigators hypothesize that patients who receive an injection of Lipogems will experience a decrease in pain of the affected knee and an increase in joint functionality in comparison to placebo. The investigators also hypothesize that patients who receive an intra-articular corticosteroid will experience decreased pain or improved functionality in the affected joint compared to placebo.

DETAILED DESCRIPTION:
Objectives:

1. The purpose of this study is to evaluate the possible benefits of reduced joint pain and increased joint functionality in patients with knee osteoarthritis after the injection of Lipogems. Based on limitations of prior research, intra-articular corticosteroids are included as a study group to be evaluated for impact on pain relief and joint functionality in comparison to placebo.
2. The investigators hypothesize that patients who receive an injection of Lipogems will experience a decrease in pain of the affected knee and an increase in joint functionality in comparison to placebo. The investigators also hypothesize that patients who receive an intra-articular corticosteroid will experience decreased pain or improved functionality in the affected joint.

Background:

Osteoarthritis (OA) causes patients considerable joint pain and leads to instability, reduced range of motion, and functional limitations. Pathologic findings of OA include decreased articular cartilage, joint space narrowing, osteophytes, subchondral sclerosis and bone cysts. Currently, treatment options are confined to symptom management only. Options for treatment include: topical preparations, nonsteroidal anti-inflammatory drugs (NSAIDs), intra-articular injections, and, in severe cases, total knee arthroplasty. Review of recent recommendations shows limitations to all available treatments. Oral NSAIDs have shown relief, but is limited to patients without risk factors or contraindications. Topical NSAIDs are recommended in elderly patients or those with GI risk factors, rather than oral NSAIDs. However, pain improvement took 12 weeks and was not long-lived, potentially due to compliance issues in application. A recent systematic review of intra-articular corticosteroids reported that, due to low-quality evidence, it is inconclusive whether intra-articular corticosteroids provided any short or long-term pain relief. Taylor's review of hyaluronic acid treatment is hampered by the variability of preparations currently on the market and shortage of double-blind placebo controlled studies, but conflicting data is reported. Osteoarthritis Research Society International currently recommends corticosteroid injections for short-term pain relief only, and is inconclusive in recommending hyaluronic acid.

The aforementioned treatment limitations have generated interest in alternative options to restore function and alleviate joint pain, some with the aim of healing damaged articular cartilage. It is well known that articular cartilage is avascular and lacks innervation, which limits its intrinsic healing and repair capabilities. Chondrocytes, derived from MSCs, have limited potential to replicate, which also limits the intrinsic healing and repair capabilities of articular cartilage. The stromal vascular fraction, containing adipose derived mesenchymal stem cells (MSCs), has historically been isolated successfully via enzymatic processes. There has been preliminary support in the literature for reduced pain and improved functional performance in patients who received MSCs as part of treatment. However, approaches to isolate MSCs are costly, time consuming, require extensive lab equipment, and are currently limited by complex regulatory issues.

Thus, interest in an alternative isolation method lead to the development of Lipogems. Lipogems is a technique to harvest, process, and inject minimally manipulated adipose tissue. This procedure is enzyme free and requires no clonal expansion or manipulation. Lipoaspirate is harvested and washed in saline solution, then processed through a closed-system device that micro-fragments the adipose tissue. This mechanical process retains the vascular architecture, mature pericytes, and MSCs for autologous injection.

As new technologies are becoming available for the treatment of OA, it is important that investigators gather high-quality data on their efficacy and outcomes. The goal of this study is to evaluate the possible benefits of reduced joint pain and increased joint functionality in patients with knee osteoarthritis after the injection of Lipogems. In addition, given the limitations of prior research on the efficacy of intra-articular corticosteroids, the investigators will also include this as an additional study group to compare to placebo. Although Lipogems is relatively new to the United States, it has been used for a variety of orthopaedic arthroscopic applications overseas including the treatment of knee OA and is being used more frequently now in the United States. As of now, there are no published studies reporting the outcomes of patients who receive Lipogems for knee OA. There have been case reports published showing favorable outcomes. Thus, this would be the first study reporting data on the efficacy of Lipogems for pain relief in knee OA in a randomized, controlled clinical trial with a larger sample of patients. It would also be the only study to date comparing Lipogems to intra-articular corticosteroids and placebo injections. The investigators feel this study design will provide new insight into the efficacy of Lipogems for pain relief of symptomatic knee OA as well as offer new data on the efficacy of intra-articular corticosteroids in this application.

ELIGIBILITY:
Inclusion Criteria:

* Age of eighteen or older
* Diagnosis of symptomatic knee osteoarthritis
* Radiographic evidence of knee osteoarthritis. Note: For the purposes of this study, radiographic evidence of knee osteoarthritis is defined as any one or more of the following: osteophytes, joint space narrowing, loss of articular cartilage thickness, subchondral sclerosis or cysts.

Exclusion Criteria:

* History of treatment with any intra-articular knee injection
* Current ligament instability as demonstrated by a positive Lachman Test, Anterior or Posterior Drawer Test, or positive Valgus or Varus Stress Test.
* Known allergy to lidocaine
* Under 18 years of age
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Richter, MD, Principal Investigator — UNM Health Sciences Center, Dept of Orthopaedic Surgery
Locations (1):
- UNM Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Background] Goldring MB, Goldring SR. Articular cartilage and subchondral bone in the pathogenesis of osteoarthritis. Ann N Y Acad Sci. 2010 Mar;1192:230-7. doi: 10.1111/j.1749-6632.2009.05240.x. PMID 20392241
- [Background] Richmond J, Hunter D, Irrgang J, Jones MH, Snyder-Mackler L, Van Durme D, Rubin C, Matzkin EG, Marx RG, Levy BA, Watters WC 3rd, Goldberg MJ, Keith M, Haralson RH 3rd, Turkelson CM, Wies JL, Anderson S, Boyer K, Sluka P, St Andre J, McGowan R; American Academy of Orthopaedic Surgeons. American Academy of Orthopaedic Surgeons clinical practice guideline on the treatment of osteoarthritis (OA) of the knee. J Bone Joint Surg Am. 2010 Apr;92(4):990-3. doi: 10.2106/JBJS.I.00982. No abstract available. PMID 20360527
- [Background] Taylor N. Nonsurgical Management of Osteoarthritis Knee Pain in the Older Adult. Clin Geriatr Med. 2017 Feb;33(1):41-51. doi: 10.1016/j.cger.2016.08.004. Epub 2016 Oct 13. PMID 27886697
- [Background] Juni P, Hari R, Rutjes AW, Fischer R, Silletta MG, Reichenbach S, da Costa BR. Intra-articular corticosteroid for knee osteoarthritis. Cochrane Database Syst Rev. 2015 Oct 22;2015(10):CD005328. doi: 10.1002/14651858.CD005328.pub3. PMID 26490760
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Sophia Fox AJ, Bedi A, Rodeo SA. The basic science of articular cartilage: structure, composition, and function. Sports Health. 2009 Nov;1(6):461-8. doi: 10.1177/1941738109350438. No abstract available. PMID 23015907
- [Background] Zlotnicki JP, Geeslin AG, Murray IR, Petrigliano FA, LaPrade RF, Mann BJ, Musahl V. Biologic Treatments for Sports Injuries II Think Tank-Current Concepts, Future Research, and Barriers to Advancement, Part 3: Articular Cartilage. Orthop J Sports Med. 2016 Apr 15;4(4):2325967116642433. doi: 10.1177/2325967116642433. eCollection 2016 Apr. PMID 27123466
- [Background] Oberbauer E, Steffenhagen C, Wurzer C, Gabriel C, Redl H, Wolbank S. Enzymatic and non-enzymatic isolation systems for adipose tissue-derived cells: current state of the art. Cell Regen. 2015 Sep 30;4:7. doi: 10.1186/s13619-015-0020-0. eCollection 2015. PMID 26435835
- [Background] Cui GH, Wang YY, Li CJ, Shi CH, Wang WS. Efficacy of mesenchymal stem cells in treating patients with osteoarthritis of the knee: A meta-analysis. Exp Ther Med. 2016 Nov;12(5):3390-3400. doi: 10.3892/etm.2016.3791. Epub 2016 Oct 11. PMID 27882169
- [Background] Pak J. Regeneration of human bones in hip osteonecrosis and human cartilage in knee osteoarthritis with autologous adipose-tissue-derived stem cells: a case series. J Med Case Rep. 2011 Jul 7;5:296. doi: 10.1186/1752-1947-5-296. PMID 21736710
- [Background] Anz AW, Hackel JG, Nilssen EC, Andrews JR. Application of biologics in the treatment of the rotator cuff, meniscus, cartilage, and osteoarthritis. J Am Acad Orthop Surg. 2014 Feb;22(2):68-79. doi: 10.5435/JAAOS-22-02-68. PMID 24486753
- [Background] Bianchi F, Maioli M, Leonardi E, Olivi E, Pasquinelli G, Valente S, Mendez AJ, Ricordi C, Raffaini M, Tremolada C, Ventura C. A new nonenzymatic method and device to obtain a fat tissue derivative highly enriched in pericyte-like elements by mild mechanical forces from human lipoaspirates. Cell Transplant. 2013;22(11):2063-77. doi: 10.3727/096368912X657855. Epub 2012 Oct 8. PMID 23051701
- [Background] Tremolada C, Colombo V, Ventura C. Adipose Tissue and Mesenchymal Stem Cells: State of the Art and Lipogems(R) Technology Development. Curr Stem Cell Rep. 2016;2(3):304-312. doi: 10.1007/s40778-016-0053-5. Epub 2016 Jul 13. PMID 27547712
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] LaPrade RF, Geeslin AG, Murray IR, Musahl V, Zlotnicki JP, Petrigliano F, Mann BJ. Biologic Treatments for Sports Injuries II Think Tank-Current Concepts, Future Research, and Barriers to Advancement, Part 1: Biologics Overview, Ligament Injury, Tendinopathy. Am J Sports Med. 2016 Dec;44(12):3270-3283. doi: 10.1177/0363546516634674. Epub 2016 Mar 29. PMID 27159318
- [Background] Deshpande BR, Katz JN, Solomon DH, Yelin EH, Hunter DJ, Messier SP, Suter LG, Losina E. Number of Persons With Symptomatic Knee Osteoarthritis in the US: Impact of Race and Ethnicity, Age, Sex, and Obesity. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1743-1750. doi: 10.1002/acr.22897. Epub 2016 Nov 3. PMID 27014966
- [Background] Losina E, Weinstein AM, Reichmann WM, Burbine SA, Solomon DH, Daigle ME, Rome BN, Chen SP, Hunter DJ, Suter LG, Jordan JM, Katz JN. Lifetime risk and age at diagnosis of symptomatic knee osteoarthritis in the US. Arthritis Care Res (Hoboken). 2013 May;65(5):703-11. doi: 10.1002/acr.21898. PMID 23203864
- [Background] Leopold SS, Redd BB, Warme WJ, Wehrle PA, Pettis PD, Shott S. Corticosteroid compared with hyaluronic acid injections for the treatment of osteoarthritis of the knee. A prospective, randomized trial. J Bone Joint Surg Am. 2003 Jul;85(7):1197-203. doi: 10.2106/00004623-200307000-00003. PMID 12851342
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Background] Wolfe F, Michaud K. Assessment of pain in rheumatoid arthritis: minimal clinically significant difference, predictors, and the effect of anti-tumor necrosis factor therapy. J Rheumatol. 2007 Aug;34(8):1674-83. Epub 2007 Jul 1. PMID 17611989
- [Background] Kim YH, Cha SM, Naidu S, Hwang WJ. Analysis of postoperative complications for superficial liposuction: a review of 2398 cases. Plast Reconstr Surg. 2011 Feb;127(2):863-871. doi: 10.1097/PRS.0b013e318200afbf. PMID 21285789
- [Background] Chow I, Alghoul MS, Khavanin N, Hanwright PJ, Mayer KE, Hume KM, Murphy RX Jr, Gutowski KA, Kim JYS. Is There a Safe Lipoaspirate Volume? A Risk Assessment Model of Liposuction Volume as a Function of Body Mass Index. Plast Reconstr Surg. 2015 Sep;136(3):474-483. doi: 10.1097/PRS.0000000000001498. PMID 26313819

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection
Started | 22 | 23 | 23
Completed | 18 | 16 | 18
Not Completed | 4 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection | Total
Number analyzed (Participants) | 22 | 23 | 23 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.8) | 56.3 (11.5) | 62.6 (8.4) | 60.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 8 | 37
  Male | 7 | 9 | 15 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Pain Scale (VAS) Over Time
Description: Scaled pain score to assess change in a patient's knee pain over time. Pain level is marked on a 100 mm line with the 0 mm corresponding to "no pain" and the 100 mm corresponding to 10/10 pain. Using a ruler, the score is determined by measuring the distance (mm) on the 100 mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Time Frame: Prior to procedure then post-procedure at 2 weeks
Measure: Median (95% Confidence Interval); unit: Median improvement in VAS pain score
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection
Number analyzed (Participants) | 22 | 23 | 23
Median improvement in VAS pain score | 1.5 [0 to 2.5] | 2.0 [0 to 5.0] | 3.0 [1.0 to 4.0]

2. Secondary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Over Time
Description: Patient self-reported outcome measure to assess pain, stiffness, and physical function in patients with knee osteoarthritis. The WOMAC consists of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The median is being reported for the three groups representing the change in the pain subscale. The following descriptors are used for all items: none, mild, moderate, severe, and extreme. These correspond to an ordinal scale of 0-4. The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. A total WOMAC score is created by summing the items for all three subscales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. The score can range from 0 to 96; however, this score is typically reported as a percentage of 100 for normalization.
Time Frame: Prior to procedure then post-procedure at 2 weeks
Measure: Median (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection
Number analyzed (Participants) | 22 | 23 | 23
scores on a scale | 3.5 [1.50 to 4.5] | 3.50 [0 to 6.5] | 5.00 [3.5 to 7]

3. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcomes Score (KOOS) Over Time
Description: Patient self-reported outcome measure to assess the patient's opinion about their knee and associated issues. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated by adding the subscales together.
Time Frame: Prior to procedure then post-procedure at 2 weeks
Measure: Median (95% Confidence Interval); unit: units on a scale in comparison to placeb
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection
Number analyzed (Participants) | 22 | 23 | 23
units on a scale in comparison to placeb | 8 [6 to 11] | 13.9 [-2.8 to 29.2] | 27.8 [19.4 to 37.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Injection | Corticosteroid Injection | Lipogems Injection
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=22) | Corticosteroid Injection (N=23) | Lipogems Injection (N=23)
Expected minor adverse event (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) — Expected mild bruising/ecchymosis and pain at abdominal fat tissue donor harvest site in all patients undergoing Lipogems procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT03379168/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT03379168/ICF_001.pdf